CLINICAL TRIAL: NCT05698615
Title: Chess Training as add-on Intervention for Adolescents With Psychiatric and Psychosomatic Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: Munich Chess academy (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-593
Record Dates: First submitted 2022-12-30; First posted 2023-01-26 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Children and Adolescents Inpatient in Psychiatric Hospital
Keywords: cognitive remediation; Chess training; working memory; decision making; executiv control; chess; cognitive change; Quality of life in adolescents

STUDY DESIGN:
Intervention Model Description: After inclusion in the study, participation in chess training begins after screening. Patients who have volunteered for chess training are then matched with patients for the comparison group. Care is taken to ensure that this group is similar to the chess group in terms of diagnoses and age ("pairwise matching").
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chess training group (Experimental): group receiving additional chess training
  Interventions: Behavioral: Chess training
- control group (No Intervention): group receiving standard therapy only

INTERVENTIONS:
Behavioral: Chess training — The chess training, which takes place as a measure for CRT with the children and adolescents, is carried out by the concept of the Munich Chess Academy. The concept applied here, "Chess according to the King's Plan", represents a holistic concept. Especially prepared for children and adolescents, theoretical aspects are illustrated in games and exercises.
  Arms: Chess training group

SUMMARY:
In the planned study, the effect of chess training on the cognitive abilities of children and adolescents with psychiatric and psychosomatic illnesses will be investigated in a naturalistic setting. Furthermore, the effects on therapy success and quality of life will be determined.Despite the thoroughly positive results, CRT has not yet been included in the official guidelines as an intervention in standard therapy; this is due, among other things, to too few studies and too little knowledge in the field of child and adolescent psychiatry. The planned study aims to fill the research gap in the field of chess training as an adjunctive intervention in children and adolescents and to provide further evidence on the relevance of CRT in child and adolescent psychiatry.

The hypotheses of the proposed study are:

1. chess training as a six-week add-on intervention will improve cognitive functioning in adolescents with psychiatric/psychosomatic disorders compared to standard treatment.
2. chess training as a six-week add-on intervention improves quality of life in adolescents with psychiatric/psychosomatic disorders compared to standard treatment.
3. chess training as a six-week add-on intervention positively influences the course of therapy in adolescents with psychiatric/psychosomatic illnesses compared to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient treatment at the Clinic for Psychiatry and Psychotherapy of Childhood and Adolescence, ZI Mannheim
* Age between 13 and 17 years
* Sufficient ability to answer questions verbally and in written form
* Ability to give consent by patients and their parents after detailed verbal and written explanation
* Consent of patients and parents must be given in paper form

Exclusion Criteria:

* Date of inpatient admission more than 3 weeks ago
* Withdrawal of informed consent
* Severe psychiatric, neurological and internal medical comorbidities

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in comorbidities | 2 time points: before and after 6 weeks chess training
  Youth Self Report (YSR, Achenbach 1991b)
Change in depressive symptoms | 2 time points: before and after 6 weeks chess training
  Beck Depression Inventory II (BDI-II, Beck, Steer, Brown 1996)
Change in anxiety symptoms | 2 time points: before and after 6 weeks chess training
  Beck Anyxiety Inventory (BAI, deutsche Version Margraf, Ehlers 2007)
Change in Quality of life | 2 time points: before and after 6 weeks chess training
  The KIDSCREEN Group Europe. (2006).
Change of the overall functional level | 2 time points: before and after 6 weeks chess training
  Global assessment of functioning (Diagnostic screening measure according to DSM-IV)
Change in mental flexibility | 2 time points: before and after 6 weeks chess training
  Dimensional Card Sorting Task (Zelazo et al., 2014
Change in attentional capacity | 2 time points: before and after 6 weeks chess training
  d2 Test of Attention (Brickenkamp 2002)
Change in Reaction inhibition | 2 time points: before and after 6 weeks chess training
  Go-No-Go Task (Sebastian et al., 2013)
Change in Fluid intelligence | 2 time points: before and after 6 weeks chess training
  Stop Signal Task (Sebastian et al., 2013)
Change in reaction time | 2 time points: before and after 6 weeks chess training
  Simple Reaction Time Task (Woods, Wyma, Yund, Herron, & Reed, 2015)

CONTACTS AND LOCATIONS:
Locations (1):
- Central Institute of Mental Health, Mannheim, Germany